CLINICAL TRIAL: NCT05150418
Title: Effects of Supplemental Oxygen on Systemic and Cerebral Hemodynamics in Experimental Hypovolemia
Brief Title: Supplemental Oxygen in Hypovolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Principal Investigator, Lars Øivind Høiseth, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1_08-06-2021
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Hypovolemia; Hyperoxia
MeSH Terms: conditions — Hypovolemia; Hyperoxia | interventions — nitrox; Air

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, crossover design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Oxygen or room air administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen (Experimental): Oxygen 15 l/min administered with face mask with reservoir.
  Interventions: Drug: Oxygen gas
- Room air (Placebo Comparator): Room air 15 l/min administered with face mask with reservoir.
  Interventions: Drug: Air

INTERVENTIONS:
Drug: Oxygen gas — Oxygen 15 l/min
  Arms: Oxygen
Drug: Air — Room air 15 l/min
  Arms: Room air

SUMMARY:
Supplemental oxygen is frequently administered in acutely and critically ill patients, specifically, it is often administered in trauma patients to avoid arterial hypoxemia and tissue hypoxia. There is also an increasing focus on potentially deleterious effects of hyperoxia. Further, the hemodynamic response to hyperoxia in hypovolemia is poorly understood.

The present study aims to investigate the effects of supplemental oxygen on systemic and cerebral hemodynamics in simulated hypovolemia in healthy volunteers.

DETAILED DESCRIPTION:
The overriding goal for the resuscitation of any critically ill patient is to ensure adequate oxygen delivery. In critically ill patients, SaO2 and PaO2 may be reduced due to lung dysfunction (e.g. atelectasis and shunt flow). Under normal circumstances, SaO2 is near to 100%, and supplemental oxygen can not increase this further. Thus, in this circumstance, providing supplemental oxygen will only increase a small, dissolved proportion. Although this proportion may be a significant fraction in some circumstances, the intention of giving supplemental oxygen is in most circumstances to ensure a high SaO2. Supplemental oxygen has been extensively used in acutely critically ill patients to avoid hypoxemia, and is recommended in severely injured trauma patients, as given by the statement: "Supplemental oxygen must be administered to all severely injured trauma patients." in the ATLS (Advanced Trauma Life Support) guidelines.

Accordingly, supplemental oxygen is often given to trauma patients, often resulting in hyperoxia. The clinical evidence for providing supplemental oxygen in all trauma patients is however scarce. The liberal use of supplemental oxygen has also largely been founded on a perception that supplemental oxygen is harmless, and that it is safer to err on the side of hyperoxia. There is however an increasing focus on possible deleterious effects of hyperoxia, especially in specific clinical circumstances. This has led to recommendations of more restrictive use of supplemental oxygen, often titrated to no more than what is necessary to achieve an adequate arterial oxygen saturation (e.g. in the range 94-98%).

In the initial treatment of trauma patients, detection and treatment of hypovolemia is of paramount importance. Hypovolemia leads to reduced cardiac filling and stroke volume. Under normal circumstances in unanesthetized humans, this is compensated by an increase in systemic vascular resistance and heart rate to maintain a normal or near-normal mean arterial pressure (MAP). At some point, these compensatory mechanisms are exhausted, and MAP typically falls abruptly.

Lower body negative pressure (LBNP) is a model of central hypovolemia where negative pressure is applied to the body from the waist-down. Thereby, blood is displaced from the central compartment of the upper body to the lower extremities and pelvis. The model has been used for more than half a century and is considered useful model for studying hypovolemia in conscious volunteers.

Normobaric hyperoxia induces vasoconstriction and reduced blood flow to several organs, including the brain, heart and skeletal muscle. One could therefore hypothesize hyperoxia leading to both an increased tolerance to hypovolemia mediated by vasoconstriction as well as a reduced tolerance mediated by reduced cerebral blood flow. One study using the LBNP-model did not find that supplemental oxygen significantly affected the hemodynamic response to simulated hypovolemia. This study did however only apply one level of LBNP and did not specifically study cerebral circulation.

Based on the above, there is a need for studies on the effects of normobaric hyperoxia on the hemodynamic response to hypovolemia. In the present study, we will study the effect of supplemental oxygen in the LBNP-model of hypovolemia in a crossover study on healthy volunteers.

In the present study, 15 healthy volunteers will be exposed to LBNP with oxygen or room air in randomized order in a crossover fashion. We will measure cardiac outout, stroke volume and middle cerebral artery blood velocity to explore effects of oxygen on these variables during hypovolemia.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Participant must be 18 years of age inclusive, at the time of signing the informed consent.
2. Participant must be under 50 years of age inclusive, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
3. Participants who are overtly healthy as determined by medical evaluation including medical history, heart and lung auscultation, focused cardiac ultrasound and measurement of cardiac conduction times.

   Sex and Contraceptive/Barrier Requirements
4. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   1. Male participants: Not applicable.
   2. Female participants:

   Use of adequate birth control for women of childbearing potential.
   * A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile when sexually active. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
   * Inclusion of WOCBP is possible when either:

     * Using at least an acceptable effective contraceptive measure (combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence). As a minimum contraception should be maintained until treatment discontinuation.

   or

   • Confirmed negative highly sensitive urine or serum pregnancy test at screening. A pregnancy test is performed at any visit before administering IMP if more than 14 days have passed since last pregnancy test. There will be no demand for post-intervention contraception.

   Informed Consent
5. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Any medical condition limiting physical exertional capacity or requiring regular medication (allergy and contraceptives excepted).
2. Pregnancy.
3. Breastfeeding.
4. History of syncope (syncope of presumed vasovagal nature with known precipitating factor excepted).
5. Any known cardiac arrhythmia. Prior/Concomitant Therapy
6. Any drug (contraceptives excepted) used on a regular basis for a chronic condition (allergy excepted).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Cardiac output | Through LBNP exposure completion, up to 35 minutes
  Cardiac output (stroke volume * heart rate)

SECONDARY OUTCOMES:
Cardiac stroke volume | Through LBNP exposure completion, up to 35 minutes
  Cardiac stroke volume as measured by suprasternal Doppler and volume-clamp method
Middle cerebral artery blood flow velocity (MCAV) | Through LBNP exposure completion, up to 35 minutes
  Middle cerebral artery blood flow velocity (MCAV) as measured by ultrasound Doppler
Time to decompensation | Through LBNP exposure completion, up to 35 minutes
  Time from start LBNP to hemodynamic decompensation

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lie SL, Hisdal J, Rehn M, Hoiseth LO. Hemodynamic effects of supplemental oxygen versus air in simulated blood loss in healthy volunteers: a randomized, controlled, double-blind, crossover trial. Intensive Care Med Exp. 2023 Nov 10;11(1):76. doi: 10.1186/s40635-023-00561-z. PMID 37947905